CLINICAL TRIAL: NCT03670277
Title: Evaluation of On-eye Optical Performances of the RMY-100 Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR-6000
Record Dates: First submitted 2018-09-12; First posted 2018-09-13 (Actual); Results first posted 2022-01-14 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Visual Acuity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- TEST arm (Experimental): For subjects enrolled in the Test arm, the Test Soft Contact Lens will be bilaterally fitted to the subject's eyes. Endpoint measures will be collected over one eye only - Test Arm: OD only.
  Interventions: Device: etafilcon A
- CONTROL arm (Experimental): Subjects enrolled in the Control Arm will be established orthokeratology lens wearers. Endpoint measures will be collected over one eye only - Control Arm: Better OK fitted eyes based on investigator's judgement.
  Interventions: Device: Habitual Orthokeratology Lenses

INTERVENTIONS:
Device: etafilcon A — Test Soft Contact Lens
  Arms: TEST arm
Device: Habitual Orthokeratology Lenses — CONTROL
  Arms: CONTROL arm

SUMMARY:
This is a two-arm parallel, non-masked, bilateral, non-dispensing study with one Test arm and one concurrent, non-randomized Control arm to evaluate the one-eye optical performances of the test soft contact lens and compare with eyes treated with orthokeratology.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. Pediatric subjects (<18 years old) must read (or be read to), understand, and sign the Statement of Information and Assent and receive a fully executed copy of the form.
  2. Adult subjects (≥18 years old) and parent(s) or legal guardian(s) of pediatric subjects must read, understand and sign the Statement of Informed Consent and receive a fully executed copy of the form.
  3. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
  4. Between 7 and 25 years of age (inclusive).
  5. Have normal eyes (i.e., no ocular medications or infections of any type).
  6. Vertex-corrected distance subjective best-sphere refraction must be between -1.00D and -5.00D (inclusive) in each eye.
  7. Cylindrical refraction must be 1.00D or less in each eye, by subjective sphero-cylindrical refraction.
  8. Have sphero-cylindrical best-corrected visual acuity of 20/25 or better in each eye.

     Below inclusion criterion is for subjects to be enrolled to the Control group only:
  9. Are existing orthokeratology patients whose current treatment has been stabilized for at least 1 months and with complete pre-treatment record, e.g., spherocylindrical refraction and corneal topography. Pre-treatment wavefront aberration measures are preferred by not required.

     Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Currently pregnant or lactating.
  2. Any systemic allergies, infectious disease (e.g., hepatitis, tuberculosis), autoimmune disease (e.g., rheumatoid arthritis), or other diseases, by self-report, which are known to interfere with contact lens wear and/or participation in the study.
  3. Use of systemic medications (e.g., chronic steroid use) that are known to interfere with contact lens wear and/or participation in the study.
  4. Any current use of ocular topical medication (occasional use of re-wetting drops is allowed).
  5. Any previous or planned ocular or intraocular surgery, including refractive surgery.
  6. Participation in any contact lens or lens care product clinical trial within 7 days prior to study enrollment.
  7. Employee or their children/relatives of investigational clinic (e.g., Investigator, Coordinator, Technician). 8 . Any ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to, aphakia, uveitis, ocular hypertension, glaucoma, severe keratoconjunctivitis sicca, history of recurrent corneal erosions, keratoconus, keratoconus suspect, pellucid marginal degeneration, entropion, ectropion, extrusions, chalazia, and recurrent styes.

  9 . Any Grade 3 or greater slit lamp findings (eg, edema, corneal neovascularization, corneal staining, tarsal abnormalities, and conjunctival injection) on the FDA scale.

  10 . Any ocular abnormality that is contraindicated contact lens wear. 11 . Any corneal scar within central 5mm 12 . Binocular vision abnormality, intermittent strabismus or strabismus. Below exclusion criteria are for subjects to be enrolled to the Test group only 13 . Current or recent (within 30 days from enrollment) rigid lens wearers. 14 . History of orthokeratology treatment. 15. Any corneal distortion resulting from ocular diseases or previous hard or rigid gas permeable contact lens wear.

Ages: 7 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2019-02-19 (Actual); Study Completion 2019-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xu Cheng, Study Chair — Johnson & Johnson Vision Care, Inc.
Locations (1):
- Centre for Ocular Research & Education, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 28 subjects were enrolled into this study at 1 clinical site. Of those enrolled, 20 subjects in the test arm were dispensed a study lens while, 8 subjects in the control arm were not dispensed, all 28 subjects who were enrolled have completed the study.
Groups:
- Test: Subjects were fit with the Test lens at Visit 2 of the study
- Control: Existing Orthokeratology patients who have >=5 mm pupil size at Visit 1 Baseline.
Period: Overall Study
Arm/Group | Test | Control
Started | 20 | 8
Completed | 20 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects dispensed a study lens
Groups:
- Total: Total of all reporting groups
Arm/Group | Test | Control | Total
Number analyzed (Participants) | 20 | 8 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.9 (3.82) | 16.8 (4.62) | 17.6 (4.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 6 | 20
  Male | 6 | 2 | 8
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 6 | 7 | 13
  White | 10 | 0 | 10
  Other | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  Canada | 20 | 8 | 28

OUTCOME MEASURES:

1. Primary Outcome: Distance Spherical Aberration (Z4, 0)
Description: Spherical aberration (Z4, 0) for a 5-mm pupil was measured by an aberrometer (COAS by AMO) with a distant viewing target at 4 m at the Baseline and post lens fitting. The Control Group only had 1 study Visit that record Baseline measurements, no intervention from the sponsor was implemented for this group, therefore data was collected on a bare eye. The Test group was fitted with the study lens at Visit 2 and data was collected with the Test lens on eye.
Time Frame: Up to Post Lens Fitting Evaluation
Population: All subjects who were administered any test article excluding subjects who dropped out prior to administering any test article. At least one observation was recorded.
Measure: Mean (Standard Deviation); unit: micron
Units Other Than Participants: Eyes
Groups:
- Test: Subjects who have >=5mm pupil size were fit with the Test lens at Visit 2 of the study
Arm/Group | Test | Control
Number analyzed (Participants) | 17 | 7
Number analyzed (Eyes) | 17 | 7
micron | 0.350 (0.066) | 0.364 (0.212)
Statistical Analysis 1: Comparison: Test vs Control; This was a pilot study for assessing the investigational test articles. As such, the sample size was not determined based on any power analysis with regard to the primary endpoint; Test type: Other — Statistically significance of difference. Statistical difference will be concluded if the lower limit was greater than 0 or the upper limit was less than 0; Mixed Models Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Least Square Mean Difference = -0.013, 95% CI 2-sided [-0.081 to 0.056], Standard Error of Mean 0.035 — Mean difference was calculated as Test - Control

2. Primary Outcome: Near Spherical Aberration (Z4, 0)
Description: Spherical aberration (Z4, 0) for a 5 mm pupil was measured by an aberrometer (COAS by AMO) with a near view target at 25 cm. at the Baseline and post lens fitting. The Control Group only had 1 study Visit that record Baseline measurements, no intervention from the sponsor was implemented for this group, therefore data was collected on a bare eye. The Test group was fitted with the study lens at Visit 2 and data was collected with the Test lens on eye.
Time Frame: Up to Post Lens Fitting Evaluation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micron
Units Other Than Participants: Eyes
Groups:
- Control: Existing Orthokeratology patients who have >=5mm pupil size at Visit1 Baseline
Arm/Group | Test | Control
Number analyzed (Participants) | 17 | 7
Number analyzed (Eyes) | 17 | 7
micron | 0.300 (0.061) | 0.272 (0.144)
Statistical Analysis 1: Comparison: Test vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Least Square Mean Difference = 0.031, 95% CI 2-sided [-0.037 to 0.100], Standard Error of Mean 0.035 — Mean difference was calculated as Test - Control

3. Secondary Outcome: Distance Off-axis Refraction at ±10°, ±20°, and ±30° Retinal Eccentricities.
Description: Distance off-axis refractions were measured by an open-field autorefractor (WAM-5500 by Grand Seiko) with distant viewing targets at 4 m and ±10°, ±20°, and ±30° off axis. at the Baseline and post lens fitting. The Control Group only had 1 study Visit that record Baseline measurements, no intervention from the sponsor was implemented for this group, therefore data was collected on a bare eye. The Test group was fitted with the study lens at Visit 2 and data was collected with the Test lens on eye.
Time Frame: Up to Post Lens Fitting Evaluation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Diopter
Units Other Than Participants: Eyes
Groups:
- Control: Existing Orthokeratology patients at Visit 1 Baseline
Arm/Group | Test | Control
Number analyzed (Participants) | 20 | 8
Number analyzed (Eyes) | 20 | 8
Diopter
  -30 | 0.3502 (3.79171) | -3.0756 (1.66232)
  -20 | -1.1344 (1.39215) | -2.4579 (1.91260)
  -10 | -0.3786 (0.94009) | -0.4444 (0.53691)
  +10 | -1.4402 (1.22240) | -1.7429 (1.16422)
  +20 | -1.9654 (1.22837) | -4.4656 (2.07377)
  +30 | -0.1098 (3.76589) | -2.5638 (2.61755)
Statistical Analysis 1: Comparison: Test vs Control; At -30°; Test type: Other — Statistically significance of difference. Statistical difference would be concluded if the lower limit was greater than 0 or the upper limit was less than 0; Mixed Models Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Least Square Mean Difference = 3.403, 95% CI 2-sided [2.557 to 4.248], Standard Error of Mean 0.431 — Mean difference was calculated as Test - Control
Statistical Analysis 2: Comparison: Test vs Control; At +30°; Test type: Other — [test comment as in outcome 3, analysis 1]; Mixed Models Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Least Square Mean Difference = 2.431, 95% CI 2-sided [1.585 to 3.277], Standard Error of Mean 0.431 — Mean difference was calculated as Test - Control

4. Secondary Outcome: Near Off-axis Refraction at ±30° Retinal Eccentricities.
Description: Near off-axis refractions were measured by an open-field autorefractor (WAM-5500 by Grand Seiko) with near viewing targets at 25 cm and ±30° off-axis. at the Baseline and post lens fitting. The Control Group only had 1 study Visit that record Baseline measurements, no intervention from the sponsor was implemented for this group, therefore data was collected on a bare eye. The Test group was fitted with the study lens at Visit 2 and data was collected with the Test lens on eye.
Time Frame: Up to Post Lens Fitting Evaluation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Diopter
Units Other Than Participants: Eyes
Arm/Group | Test | Control
Number analyzed (Participants) | 20 | 8
Number analyzed (Eyes) | 20 | 8
Diopter
  -30 | -2.3463 (3.13560) | -5.3558 (2.49516)
  +30 | -3.6046 (3.37323) | -4.9883 (3.77839)
Statistical Analysis 1: Comparison: Test vs Control; At -30°; Test type: Other — [test comment as in outcome 3, analysis 1]; Mixed Models Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Least Square Mean Difference = 3.039, 95% CI 2-sided [1.854 to 4.225], Standard Error of Mean 0.603 — Mean Difference was calculated as Test - Control
Statistical Analysis 2: Comparison: Test vs Control; At +30°; Test type: Other — [test comment as in outcome 3, analysis 1]; Mixed Models Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Least Square Mean Difference = 1.414, 95% CI 2-sided [0.228 to 2.599], Standard Error of Mean 0.603 — Mean Difference was calculated as Test - Control

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study; approximately 2 days up to 10 days.
Arm/Group | Test | Control
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/8
Other Adverse Events (participants affected / at risk) | 0/20 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-05): https://cdn.clinicaltrials.gov/large-docs/77/NCT03670277/Prot_SAP_000.pdf